CLINICAL TRIAL: NCT03868475
Title: Efficacy, Safety, Cosmesis and Patient Satisfaction With Vacuum-Assisted Percutaneous Excision (VAPE) Compared With Standard Surgical Excision (X) of Non-malignant, Borderline or High-risk Breast Lesions: A Randomized Controlled Trial
Brief Title: Comparing Vacuum-Assisted Percutaneous Excision to Open Surgical Excision for Borderline or High-Risk Breast Lesions
Acronym: VAPEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Muriel Brackstone, Associate Professor of Surgery & Oncology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Breast Fibroadenoma; Atypical Ductal Hyperplasia; Atypical Lobular Hyperplasia; Lobular Carcinoma in Situ; Flat Epithelial Atypia; Phyllodes; Fibroadenoma; Phyllodes Breast Tumor; Radial Scar; Breast Papilloma; Complex Sclerosing Papillary Lesion of the Breast
Keywords: High-risk breast lesions; Vacuum-assisted excision; Vacuum-assisted biopsy; Surgical excisional biopsy; Complete removal; Patient satisfaction; Cosmesis
MeSH Terms: conditions — Fibroadenoma; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Phyllodes Tumor; Cicatrix; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vacuum-assisted percutaneous excision (Experimental): Patients will undergo vacuum-assisted percutaneous excision (VAPE). The intervention group will have post-procedure imaging the same day to confirm complete excision.
  The intervention group will then have imaging at 6, 12, and 24 months as per the radiology algorithms for following suspicious lesions (BIRADS 3 category). If at any point during the imaging follow up, a suspicious lesion or calcifications are detected, it would be sampled with core needle biopsy and then surgically excised as appropriate.
  The intervention group will also be seen in clinic at 1 month with no imaging and then at 6, 12, and 24 months to correspond to the imaging visits.
  Interventions: Procedure: Vacuum-assisted percutaneous excision
- Open surgical excision (Active Comparator): Patients will undergo standard open surgical excision.
  The control group will then have follow up imaging at 12 and 24 months as per the usual radiology algorithms following excision of a lesion. If at any point during the imaging follow up, a suspicious lesion or calcifications are detected, it would be sampled with core needle biopsy and then surgically excised as appropriate.
  The control group will also be seen in clinic at 1 month with no imaging and then at 12 and 24 months to correspond to the imaging visits.
  Interventions: Procedure: Open surgical excision

INTERVENTIONS:
Procedure: Vacuum-assisted percutaneous excision — The intervention group will undergo the vacuum assisted percutaneous excision (VAPE). All VAPE procedures will be performed on a digital supine table using the ATEC© Breast Biopsy System hand piece (Hologic) with a 9-gauge needle and a 10 or 20 mm aperture providing 6-mmHg of suction strength to completely excise the breast lesion.
  Arms: Vacuum-assisted percutaneous excision
Procedure: Open surgical excision — The control group will undergo standard open surgical excision of the breast lesion. This will be done in the operating room using preoperative image-guided localization with radioactive seed (I-125) or in the procedure room of the Breast Care Centre if appropriate (i.e. lesion is palpable and localization is not required).
  Arms: Open surgical excision

SUMMARY:
This randomized controlled trial compares vacuum-assisted percutaneous excision to open standard surgical excision in women who have high-risk or borderline, non-malignant breast lesions with respect to efficacy, safety, cosmesis and patient satisfaction.

DETAILED DESCRIPTION:
In women diagnosed with high-risk or borderline, non-malignant breast lesions, is vacuum-assisted percutaneous excision (VAPE) comparable to open standard surgical excision with respect to efficacy, safety, cosmesis and patient satisfaction?

With the increase in breast imaging for screening there has been corresponding rise in detection of high-risk/borderline, non-malignant breast lesions that require surgical excision to confirm diagnosis and rule out underlying malignancy. Image-guided vacuum-assisted percutaneous excision (VAPE) could offer an alternative to standard open surgical excision for complete excision of these lesions with a possible improvement in patient satisfaction and cosmetic outcomes and decreased complications.

In this single-centre, non-inferiority designed prospective randomized, open label controlled trial, women over 18 years who are found to have a borderline or high-risk, non-malignant breast lesions on core needle biopsy will be considered eligible. Exclusion criteria will be women with a greater than 25% lifetime risk of breast cancer, patients whose pathology and imaging are discordant, and those with extensive calcifications extending over 2cm, a mass larger than 2 cm, or lesions with high-risk features. Informed consent will be obtained and patients will be randomized to standard surgical excision or VAPE. They will then be followed with imaging as appropriate.

The primary outcome measure is the incidence of complete removal of the lesion. The secondary outcome measures are patient satisfaction, cosmetic outcomes and complications such as bleeding and infection.

This trial is the first randomized controlled trial to investigate the role of VAPE compared to standard surgical excision as a means of completely excising borderline or high-risk breast, non-malignant breast lesions. The investigators hypothesize that VAPE will show comparable efficacy and may even have improved safety, cosmesis and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Women over age 18 with a core biopsy proven borderline or high-risk breast lesion that requires further excision for management based on the surgeon's assessment
* Informed consent must be obtained.

Exclusion Criteria:

* Women who are considered high-risk based on a greater than 25% lifetime risk of breast cancer as per the IBIS (International Breast Cancer Intervention Study) Breast Cancer Risk Evaluation Tool
* Pathology that is felt to be discordant with imaging
* Extensive calcifications extending more than 20 mm and/or masses greater than 30 mm
* The following lesions will be excluded based on their increased risk of upstaging; lesions (other than fibroadenomas, phyllodes and papillomas) that are associated with a palpable mass, ADH (atypical ductal hyperplasia) with high-risk features (ADH with zonal necrosis, significant cytological atypia or more than 2 foci), LCIS (lobular carcinoma in situ) with high-risk features (associated with ADH, pleomorphic LCIS, zonal necrosis and > 4 foci) or discordant with imaging, papilloma with atypia, and spindle cell lesion (especially if there is atypia).
* Lesions that are suspicious for borderline or malignant Phyllodes, DCIS (ductal carcinoma in situ), invasive mammary carcinoma, or encapsulated papillary carcinoma
* Any lesion that either the radiologist, pathologist or surgeon feels is not amenable to VAPE or surgical excision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete removal of the breast lesion | 24 months
  No evidence of residual lesion at the time of excision or on follow up imaging exams and no need for further surgical re-excision for residual lesion.

SECONDARY OUTCOMES:
Patient satisfaction | 12 months
  Patient satisfaction as assessed by the BREAST-Q questionnaire for breast conserving therapy, Version 2.0, a validated patient-reported outcome measure that quantifies health-related quality of life and patient satisfaction. It will be completed preoperatively, and at 1, 6, and 12 months postoperatively.
  There are three components being assessed:
  1. Physical well-being: 10 items scored using a 3-point scale (1=none of the time, 2=some of the time, 3=all of the time).
  2. Psychosocial well-being: 10 items scored using a 5-point scale (1=none of the time, 2=a little of the time, 3=some of the time, 4=most of the time, 5=all of the time).
  3. Satisfaction with breasts: 4 items scored using a 4-point scale (1=very dissatisfied, 2=somewhat dissatisfied, 3=somewhat satisfied, 4=very satisfied).
  Each component has a raw scale summed score (the sum of all the scores for each item) that is converted into a score from 0 (worst) to 100 (best) for analysis.
Cosmesis | 12 months
  Cosmesis as assessed by the Modified Harvard-Harris Cosmetic Scale, a validated four-point scale that describes the overall aesthetic appearance of the breasts (categorical scale = excellent, good, fair or poor). It will be administered to both the patients as a self-assessment and the surgeons before the intervention and at various time points postoperatively (1 month, 6 months, and 12 months).

OTHER OUTCOMES:
Rate of Surgical Site Infections (SSI) | 30 days
  As defined by the Center for Disease Control and Prevention (CDC) criteria (Pearson) as infection occurring within the first 30 post-operative days with at least one of the following: (a) purulent drainage from the incision or biopsy site, (b) organisms isolated from an aseptically obtained culture of fluid or tissue, (c) incision is deliberately opened by a surgeon AND patient has at least one of the following signs or symptoms: pain or tenderness, localized swelling, erythema, or heat, or (d) diagnosis of SSI by the surgeon
Number of patients that have a post-procedural bleeding or hematoma | 30 days
  Any bleeding or hematoma that requires an intervention (such as re-operation to evacuate the hematoma or control the bleeding or aspiration of the hematoma)

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Brackstone, PhD, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's

IPD SHARING:
Plan to Share IPD: No